CLINICAL TRIAL: NCT00875940
Title: Right Ventricular Hypertrophy and Pulmonary Hypertension: A Correlation Analysis Between Tc-99m Tetrofosmin SPECT Adn Echocardiography
Brief Title: Right Ventricular Hypertrophy and Pulmonary Hypertension: A Correlation Analysis
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Responsible Party: Myron Gerson M.D., University Internal Medicine Associates
Other Study IDs: IRB # 08-01-24-02
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2009-04-06 (Estimated); Status verified 2009-04

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1: Patients having both Tc-99m perfusion scan and echocardiogram.
  Interventions: Other: Diagnostic imaging procedures.

INTERVENTIONS:
Other: Diagnostic imaging procedures.

SUMMARY:
The study hypothesis is that a quantitative index can be derived from Tc-99m myocardial perfusion scans that accurately identifies the presence of left ventricular hypertrophy and pulmonary hypertension. Echocardiography provides the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Must have an interpretable Tc-99m myocardial perfusion scan and an interpretable echocardiogram.

Exclusion Criteria:

* Technically inadequate noninvasive test.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hospital population having diagnostic testing.
Sampling Method: Non-Probability Sample
Dates: Start 2008-02; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of quantitation of Tc-99m perfusion scans for identification of pulmonary hypertension. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States